CLINICAL TRIAL: NCT05561517
Title: Competition Induced Hyperglycemia in Athletes With Type 1 Diabetes
Acronym: EXCITE-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 94654
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes; Hyperglycemia Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 12 athletes with T1D and 12 healthy athletes are included in a prospective experimental randomized, cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Competition (Active Comparator): Participation in a 5 K competition (running)
  Interventions: Other: 5 K running
- Training (Active Comparator): Performing a 5 K up-tempo training bout (running)
  Interventions: Other: 5 K running

INTERVENTIONS:
Other: 5 K running — The 5 K running competition will induce increased stress levels and thereby lead to increased levels of hyperglycemia.

SUMMARY:
Design and methods 12 athletes with T1D and 12 healthy athletes are included in a prospective experimental randomized, cross-over study. Athletes are provided with a Dexcom G6 CGM to measure glucose excursions before, during and after exercise and a Holter ECG-E-patch to measure HRV. Psychological stress levels are assessed from Competitive State Anxiety Inventory-2.

The athletes are studied on two occasions: Day 1: 5K running competition and Day 2: 5K high intensity training session (running) in the athletes' regular training environment.

Endpoints Primary endpoints: Change in plasma glucose from start of exercise to end of exercise during competition compared to training.

Secondary endpoints: Hormonal response (cortisol, adrenalin, noradrenaline). Changes in heart rate and HRV before, during and after exercise. CGM-glucose and plasma glucose discrepancies.

DETAILED DESCRIPTION:
Design 12 athletes with T1D and 12 healthy athletes are included in a prospective experimental randomized, cross-over study.

Screening visit Investigator Rakel Fuglsang Johansen will orally inform eligible athletes about the study at the screening visit at Steno Diabetes Center Aarhus. Individuals who have agreed to join the study (given oral and written informed consent), will have a short physically examination performed including measurement of blood pressure, height, weight, and heart and lung auscultation and screening blood samples (kidney, liver, and blood counts, lipids, and HbA1c) will be taken.

Prior to study days Within 1 month prior to the 1st study day, eligible participants will also be invited to perform a maximal incremental test to volitional exhaustion to determine their individual VO2 max. The test will be performed on a treadmill.

The athletes come to the outpatient clinic 2 days prior to the 1st study day (training or competition), where they are provided with a Dexcom G6 CGM to measure glucose excursions before, during and after exercise and a Holter ECG-E-patch to measure HRV. Instructions on food and liquid intake prior to study days are provided.

The participants are required to refrain from any intense or prolonged physical activity and alcohol consumption 48 hours prior to study days and instructed to consume a weight maintaining diet according to recommended guidelines (approx. 20 % fat, 30 % protein and 50 % carbohydrate). The participants are asked to keep a food diary and to match their food intake as accurate as possible before the two study days.

Participants with T1D should not change their insulin treatment or strategies prior to or during the study days. If the participant has experienced severe hypoglycemia (glucose measurement below 2.8 mmol/L) within 24 h hours before the study day, a new study day will be arranged. This in order to avoid that upstream hypoglycemia will affect the glucoregulatory responses during the study day, and because of the increased risk of a new hypoglycemic events.

Study days The athletes participate in a competition day and a training day in randomized order.

On the competition day, the athletes participate in a 5 km race. The last meal must be consumed at least 2 hours before the competition and the athlete is not allowed to consume anything until 1 hour after the completion of the competition, where the last blood sample will be taken. Participants with T1D should adhere to the same fasting period, but if this is not possible due to hypoglycemia, then the type and amount of food/fluid intake is recorded.

Twenty minutes before the start of the competition the initial blood samples are taken. After the athlete has completed the competition, blood sampling is repeated after 10, 20, 30, and 60 minutes. At each time point, blood samples for measurement of hormonal response (cortisol, adrenalin, noradrenaline, glucagon, insulin, growth hormone) and circulating metabolites (glucose, free fatty acids, glycerol, triglyceride, lactate) are collected. During this period, the athlete is interviewed about dietary intake within the last 24 hours and psychological stress in assessed by use of the Competitive State Anxiety Inventory-2 (SCAI-2) questionnaire. After the last blood sample has been taken, the athlete is allowed to eat and drink as usual, and the study day is completed.

On the training day, the athletes perform a 5 km high-intensity training run, but in the athletes' regular training environment without the element of competition. The time to complete the 5 km is recorded. The training sessions are performed at the same time of the day as on the competition day and the same rules apply as on the competition day regarding food and beverage intake. Blood samples are collected in the same manner as on the competition day. Once again, an interview regarding food intake and stress level is performed.

The competition day and the training day are performed three to six days apart. During the 10-day period where the CGM device is worn, data are recorded in a personal study diary listing start and end of training sessions. Food intake is recorded in the diary 24 prior to and during the study day, as well as hypoglycemic events within this period.

ELIGIBILITY:
Inclusion Criteria:

* T1D and healthy athletes who are otherwise healthy
* Age between 18 and 65 years
* HbA1c less than 70 mmol/mol
* The athletes must be engaged in competitive sports that includes running, and agree to participate in a local 5 km running competition within 3 months

Exclusion Criteria:

* Proliferative retinopathy
* Hypoglycemia unawareness
* Heart disease and other conditions which may be negatively affected by the VO2 max test and study days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | Plasma glucose is measured Twenty minutes before the start of the competition until 60 minutes after the competition.
  Change in plasma glucose from start of exercise to end of exercise during competition compared to training. Level of plasma glucose at the beginning and end of competition versus training session.

CONTACTS AND LOCATIONS:
Overall Officials: Esben Soendergaard, Principal Investigator — University of Aarhus
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No